CLINICAL TRIAL: NCT04021173
Title: A Multicenter, Randomized, Double-blind, Placebo-parallel, Phase II Clinical Trial of the Efficacy and Safety of Anfibatide in Treating Patients With Acquired Thrombotic Thrombocytopenic Purpura (TTP)
Brief Title: A Clinical Study of Anfibatide in Acquired Thrombotic Thrombocytopenic Purpura (TTP)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APT-ZK-201901
Record Dates: First submitted 2019-07-15; First posted 2019-07-16 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Acquired Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — agkisacucetin protein, Agkistrodon acutus; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anfibatide (Experimental)
  Interventions: Drug: Anfibatide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Anfibatide — 5 IU/60kg intravenous infusion follow by 0.002 IU/kg/h continuous intravenous infusion
  Other Names: Anti-platelet thrombolysin for injection
  Arms: Anfibatide
Drug: Placebos — 5 IU/60kg intravenous infusion follow by 0.002 IU/kg/h continuous intravenous infusion
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, parallel, placebo-controlled phase II clinical study. It is planned to recruit 74 patients with acquired thrombotic thrombocytopenic purpura (TTP). To evaluate the efficacy and safety of Anfibatide as an adjuvant therapy for plasma exchange in patients with acquired TTP.

DETAILED DESCRIPTION:
The study will consist of 3 periods: screening(up to 7 days), treatment and follow-up(up to 3 months). Subjects are assigned in a 1:1 ratio to Anfibatide or placebo during plasma exchange with the use of a computerized randomization schedule. The administration is 5 IU/60kg intravenous infusion and 0.002 IU/kg/h continuous intravenous infusion. Plasma exchange as the main treatment method is performed daily on the 5th day of solstice and then adjusted to every other day. Fresh frozen plasma（FFP）and cryoprecipitate-reduced plasma are preferred. Subjects will receive the study drug immediately after daily plasma exchange.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male subjects with 18 years of age or older.
2. Subjects with diagnosis of TTP.
3. Necessitating plasma exchange.
4. Obtained, signed and dated informed consent.

Exclusion Criteria:

1. Platelet count greater or equal to 100*10^9/μL.
2. Severe heart, liver and kidney dysfunction, including those with glutamic-pyruvic transaminase ≥ 5xULN，glomerular filtration rate <30ml/min.
3. Uncontrolled severe active infection.
4. Known congenital TTP.
5. Subjects with malignant tumors in the past 5 years.
6. Other diseases that cause microangiopathy hemolytic anemia and thrombocytopenia, such as disseminated intravascular coagulation (DIC), antiphospholipid antibody syndrome, hemolytic uremic syndrome, malignant hypertension, and transplant-related microangiopathy.
7. Pregnant or lactating women. Subjects of reproductive age, are unable to use effective contraceptive methods during the study period.
8. Severe active bleeding or progressive aggravation of bleeding symptoms.
9. Subjects who have received plasmapheresis during the treatment of the onset of the disease.
10. Subject is participating in other clinical stuy or is less than 3 months away from the end of previous clinical study.
11. Subject who have participated in other clinical trials related to Anfibatide.
12. Severe or life threatening clinical condition other than TTP that would impair participation in the trial.
13. Life expectation less than 1 week.
14. Known to be allergic to the drugs or ingredients in the study.
15. Inability to follow programme requirements and procedures.
16. Subjects who are not eligible to participate in this clinical study as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Time to response of treatment | up to 21days
  Time to response of treatment ,defined by a recovery of platelets ≥100*10^9/l

SECONDARY OUTCOMES:
Remission rate | up to 21days
  Number of subjects with remission

OTHER OUTCOMES:
Complete remission rate | up to 21 days
  Number of subjects with complete remission
Number of plasma exchange | up to 21 days
  The number of plasma exchange to achieved remission.
Volume of plasma | up to 21 days
  The volume of plasma to achieved remission.
Time to achieve threshold values of biological markers. | up to 3 months
  The biological markers include platelets，LDH and creatinine.
Total mortality | up to 21days and the ensuing 30 days
  Total mortality within the plasma exchange treatment period and the ensuing 30 days.
Number of exacerbations of TTP and time to first exacerbation of TTP. | up to 1 month
  Exacerbation is defined as recurrent thrombocytopenia following a response and requiring a reinitiation of daily plasma exchange treatment after ≥ 1 day but ≤ 30 days of no plasma exchange treatment.
Number of subjects relapsing of TTP for maximum of 3 months and time to first relapse of TTP. | up to 3 months
  Relapse is defined as novo event of TTP that occurs later than 30 days after the last plasma exchange.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, MD, Study Director — Shanghai Ruijing Hospital
Locations (1):
- Shanghai Ruijing Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No